CLINICAL TRIAL: NCT06573190
Title: The Value of Fibroscan® in Assessing the Liver Status and Presence of MASLD/MASH in Patients With Chronic Hepatitis B and Monitoring Changes by Antiviral Therapy: Faraday Study
Brief Title: Liver Status and Presence of MASLD/MASH in Patients With Chronic Hepatitis B
Acronym: Faraday
Status: Completed | Type: Observational
Sponsor: Yaşar Bayındır, MD (Other)
Collaborators: Nobel Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Yaşar Bayındır, MD, Chief Physician, Prof. Dr., M.D., Guven Health Group
Organization: Guven Health Group (Other)
Other Study IDs: Guven Health Group Faraday
Record Dates: First submitted 2024-08-07; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Chronic Hepatitis B; Hepatic Steatosis
Keywords: Chronic hepatitis B; Metabolic syndrome; Hepatic fibrosis; Hepatic steatosis
MeSH Terms: conditions — Hepatitis B, Chronic; Fatty Liver; Metabolic Syndrome; Liver Cirrhosis | interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy materials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic hepatitis B patients: Patients aged 18 years and older with HBsAg positivity for more than six months and HBV-DNA level >2,000 IU/ml
  Interventions: Diagnostic Test: Transient elastography; Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Diagnostic Test: Transient elastography — Liver Stiffness Measurement, Controlled Attenuation Parameter
  Other Names: Fibroscan
Drug: Tenofovir Disoproxil Fumarate — Guided Therapy
  Other Names: TDF

SUMMARY:
The aim of the study was to evaluate the consistency between liver biopsy and Liver Stiffness Measurement (LSM) for fibrosis and controlled attenuation parameter (CAP) for steatosis in FibroScan® in patients with chronic hepatitis B. The secondary aim of the study was to demonstrate the efficacy of FibroScan® for following the CHB patients at 12th month of antiviral therapy.

The study was prospectively planned in four different centers. Patients with HBsAg positivity for more than six months and HBV-DNA>2,000 IU/mL, underwent liver biopsy and FibroScan® together within two week. FibroScan® was performed twice, before the antiviral therapy and one year later.

DETAILED DESCRIPTION:
Patients aged 18 years and older with HBsAg positivity for more than six months and HBV-DNA level >2,000 IU/ml were included in the study. The exclusion criteria were established as presence of cirrhosis, alcohol consumption >140 g/week for women and 210 g/week for men, hepatitis C, hepatitis D and/or HIV coinfections.

The baseline characteristics including patient demographics, BMI, comorbidities, LSM and CAP via transient elastography (FibroScan®), liver ultrasound, HBV serology, platelet count, ALT, HBV viral load.

All patients underwent liver biopsy before initiating antiviral therapy, with a maximum interval of two week between liver biopsy and the FibroScan®.

Transient elastography was performed by a certified operator, using the M probe for patients with skin to capsule distance < 2.5 cm or an XL probe for patients with skin to capsule distance > 2.5 cm. Patients were fasted for > 2 h before FibroScan®. At least 10 successful measurements were performed and recorded.

Fibrosis stage by Liver Stiffness Measurement (LSM) and steatosis by Controlled Attenuation Parameter (CAP) were investigated on FibroScan® for MASLD and MASH. Obese or diabetic patients with a CAP value >240 dB/m were considered MASLD. Patients with normal BMI and nondiabetic patients had at least two risk factors for metabolic dysfunction were also considered to have MASLD. Patients with MASLD and concomitant necroinflammation in the liver were considered as MASH. Necroinflammation was considered as LSM ≥7.2 kPa in patients with MASLD or LSM >5.5 kPa in patients with liver injury (histologic and/or ALT>NSU).

The study protocol was approved by the Ethics Committee of Dicle University (Protocol number: 2022/261) The IBM SPSS 21.0 statistical software for Windows was used for the statistical evaluation of the research data. The measurable variables were presented as the mean ± standard deviation (SD), while the categorical variables were presented as the number and percentage (%). Spearman's rho correlation analysis was performed to determine the relationship between the variables. The hypotheses were bidirectional, and p ≤0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older with HBsAg positivity for more than six months
* Patients have HBV-DNA level >2,000 IU/ml for more than six months

Exclusion Criteria:

* Presence of cirrhosis
* Alcohol consumption >140 g/week in women and 210 g/week in men
* Hepatitis C coinfection
* Hepatitis D and/or HIV coinfections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older with HBsAg positivity for more than six months and HBV-DNA level >2,000 IU/ml were included in the study. The exclusion criteria were established as presence of cirrhosis, alcohol consumption >140 g/week for women and 210 g/week for men, hepatitis C, hepatitis D and/or HIV coinfections.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Histological activity index (HAI) evaluatin by liver biopsy in patients with chronic hepatitis B before initiating antiviral therapy. | 23.01.2023-25.04.2023
  All patients underwent liver biopsy before initiating antiviral therapy, for evaluating histological activity index (HAI). According to modified HAI system (Ishak), HAI scores ranging from 0 to 18 were used.
Fibrosis score evaluation by liver biopsy in patients with chronic hepatitis B before initiating antiviral therapy. | 23.01.2023-25.04.2023
  All patients underwent liver biopsy before initiating antiviral therapy, for evaluating fibrosis score. According to modified HAI system (Ishak), seven point scale ranging from 0 to 6 for fibrosis stage.
Hepatic steatosis evaluation by Controlled Attenuation Parameter (CAP) on FibroScan® in patients with chronic hepatitis B before initiating antiviral therapy. | 23.01.2023-25.04.2023
  FibroScan® measurements were perfomred at most two weeks apart from biopsy. Hepatic steatosis by Controlled Attenuation Parameter (CAP) were investigated on FibroScan® for MASLD and MASH. Obese or diabetic patients with a CAP value >240 dB/m were considered MASLD. Patients with normal BMI and nondiabetic patients had at least two risk factors for metabolic dysfunction were also considered to have MASLD.
Fibrosis stage by Liver Stiffness Measurement (LSM) on FibroScan® in patients with chronic hepatitis B before initiating antiviral therapy. | 23.01.2023-25.04.2023
  FibroScan® measurements were perfomred at most two weeks apart from biopsy. Fibrosis stage by Liver Stiffness Measurement (LSM) was investigated on FibroScan®. Necroinflammation was considered as LSM ≥7.2 kPa in patients with MASLD. Patients with MASLD and concomitant necroinflammation in the liver were considered as MASH.

SECONDARY OUTCOMES:
Hepatic steatosis evaluation by Controlled Attenuation Parameter (CAP) on FibroScan® in patients with chronic hepatitis B at 12th month of antiviral therapy. | 23.01.2024-25.04.2024
  Hepatic steatosis by Controlled Attenuation Parameter (CAP) were investigated on FibroScan® for MASLD and MASH. Obese or diabetic patients with a CAP value >240 dB/m were considered MASLD. Patients with normal BMI and nondiabetic patients had at least two risk factors for metabolic dysfunction were also considered to have MASLD.
Fibrosis stage by Liver Stiffness Measurement (LSM) on FibroScan® in patients with chronic hepatitis B. | 23.01.2024-25.04.2024
  FibroScan® measurements were performed at most two weeks apart from biopsy. Fibrosis stage by Liver Stiffness Measurement (LSM) was investigated on FibroScan®. Necroinflammation was considered as LSM ≥7.2 kPa in patients with MASLD. Patients with MASLD and concomitant necroinflammation in the liver were considered as MASH.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kemal Çelen, MD, Principal Investigator — Dicle University, Medical Faculty, Department of Infectious Diseases
Locations (1):
- Guven Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vittal A, Ghany MG. WHO Guidelines for Prevention, Care and Treatment of Individuals Infected with HBV: A US Perspective. Clin Liver Dis. 2019 Aug;23(3):417-432. doi: 10.1016/j.cld.2019.04.008. PMID 31266617
- [Result] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Result] Wang L, Wang Y, Liu S, Zhai X, Zhou G, Lu F, Zhao J. Nonalcoholic fatty liver disease is associated with lower hepatitis B viral load and antiviral response in pediatric population. J Gastroenterol. 2019 Dec;54(12):1096-1105. doi: 10.1007/s00535-019-01594-6. Epub 2019 May 27. PMID 31134334
- [Result] Jiang K, Zhang L, Li J, Hu H, Huang Q, Qiu T, Mo X, Ren J, Guo W, Tao Y, Cui H, Zuo Y, Chen X, Xie Y, Li Y, Liang H, Liu Z, Xie L, Mao R, Jiang Q, Huang K. Diagnostic efficacy of FibroScan for liver inflammation in patients with chronic hepatitis B: a single-center study with 1185 liver biopsies as controls. BMC Gastroenterol. 2022 Jan 29;22(1):37. doi: 10.1186/s12876-022-02108-0. PMID 35090390

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT06573190/Prot_SAP_000.pdf